CLINICAL TRIAL: NCT06499493
Title: Effects of Myofascial Induction Pressure Pain Threshold in Trigger Points of the Proximal Muscles of Gastrocnemius: A Prepost Study
Brief Title: Effects of Myofascial Induction Pressure Pain Threshold in Trigger Points of the Proximal Muscles of Gastrocnemius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Physiotherapist responsible area, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2911202021420B
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Myofascial Trigger Point; Gastrocnemius Muscle; Manual Therapy; Pain Threshold
Keywords: gastrocnemius muscle; range of motion; lower limb; therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Myofascial induction in gastrocnemius (Experimental): A 3-pass shallow leg gliding technique was applied first, followed by 5 minutes of the deep myofascial calf induction technique described by Pilat.
  Interventions: Other: Myofascial induction in gastrocnemius muscle

INTERVENTIONS:
Other: Myofascial induction in gastrocnemius muscle — A 3-pass shallow leg gliding technique was applied first, followed by 5 minutes of the deep myofascial calf induction technique described by Pilat.

SUMMARY:
In the present study we will test the effects of myofascial induction technique in the muscles close to the application in the gastrocnemius muscle.

DETAILED DESCRIPTION:
In the present study we will test the effects of myofascial induction technique on nearby muscles. The calf maneuver proposed by Pilat for myofascial induction will be applied and the effects on the pain pressure threshold of the trigger points of the flexor digitorum brevis biceps femoris extensor digitorum longus muscles will be observed.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged 18-39 years.
* Healthy subjects with trigger point 1 of the gastrocnemius muscle in both lower limbs.

Exclusion criteria;

* Diagnosis of lower limb injury, including any tendinopathy, bursitis, ligamentous involvement and/or fasciitis.
* History of lower limb surgery or history of lower limb injury with residual symptoms (pain or sensation of sensation) within the last year.
* Participants could not have undergone ankle stretching or any other treatment.
* Diabetes due to possible impaired distal arterial circulation.
* Foot deformity, cavus and flat feet.
* Foot deformities such as hammertoes and hallux valgus,
* plantar calluses.
* Dysfunction of the lower extremities or chronic injuries.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
1.Pressure pain threshold in flexor digitorum brevis, biceps femoris, extensor digitorum brevis muscles before intervention | Immediately before intervention.
  The pressure at which the patient begins to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons.
2.Pressure pain threshold in flexor digitorum brevis, biceps femoris, extensor digitorum brevis muscles after intervention | Immediately after the intervention.
  The joint range is measured in dorsiflexion of the ankle joint with the knee extended under load and is measured with an inclinometer in degrees.Measured in grades.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No